CLINICAL TRIAL: NCT07063992
Title: Effects of Thoracic Spine Manipulation With and Without Costovertebral Joint Manipulation in Patients With Non-specific Mid-back Pain
Brief Title: Effects of Thoracic Spine Manipulation With and Without Costovertebral Joint Manipulation in Patients Mid-back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0142 Alishah
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Back Pain
Keywords: Craniovertebral Angle; Mid-Back Pain; muscle strength
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thoracic facet manipulations (Experimental): Group A will receive thoracic facet manipulations of the restricted segments between T3 to T9, in the prone position and cephalic direction. The duration of the intervention will be followed by 4 weeks 3 sessions each week and pre- and post-intervention observations will be recorded.
  * Bilateral hypothenar
  * Cross bilateral hypothenar manipulation
  Interventions: Other: thoracic facet manipulations
- thoracic facet and costovertebral manipulations (Experimental): Group B will receive thoracic facet and costovertebral manipulations of the restricted segments between T3 to T9 and ribs 3 to 9 (costovertebral joints), in the prone position. The duration of the intervention will be followed by 4 weeks 3 sessions each week and pre and post-intervention observations will be recorded.
  * Hypothenar Costal Manipulative technique
  * Ilial Hypothenar costal manipulation between T3-T9
  Interventions: Other: thoracic facet and costovertebral manipulations

INTERVENTIONS:
Other: thoracic facet manipulations — Group A will receive thoracic facet manipulations of the restricted segments between T3 to T9, in the prone position and cephalic direction. The duration of the intervention will be followed by 4 weeks 3 sessions each week and pre- and post-intervention observations will be recorded.
  Bilateral hypothenar Cross bilateral hypothenar manipulationThese flexibility exercises will be targeted for
  * Rhomboid and middle trapezius stretching (2-3 times daily; 3 sets for 30 seconds))
  * Pectoralis muscle stretch in a corner (2-3 times daily; 3 sets for 30 seconds)
  * Prone on the elbow with upper thoracic extension exercise (2-3 times daily; 3 sets for 30 seconds) .
  The postural exercises will be the following
  * Postural strengthening/ stabilization with back to a wall. The participant will press their arms into the wall while retracting scapulae.
  * Trunk rotation stretching in the sitting position
  Arms: thoracic facet manipulations
Other: thoracic facet and costovertebral manipulations — Group B will receive thoracic facet and costovertebral manipulations of the restricted segments between T3 to T9 and ribs 3 to 9 (costovertebral joints), in the prone position. The duration of the intervention will be followed by 4 weeks 3 sessions each week and pre and post-intervention observations will be recorded.
  Hypothenar Costal Manipulative technique Ilial Hypothenar costal manipulation between T3-T9
  Arms: thoracic facet and costovertebral manipulations

SUMMARY:
Mid-back pain (mbp) is defined as pain occurring within the limits of the third thoracic (T3) and ninth thoracic (T9) vertebrae, caused by the dysfunction of the musculoskeletal structures in the thoracic spine. It can present as pain and/or burning between the shoulder blades with reduced thoracic spine mobility and increased muscle tension. Congenital disorders such as scoliosis and Scheuermann's disease, or acquired disorders such as thoracic facet and costovertebral joint dysfunction may cause mid back pain.

DETAILED DESCRIPTION:
Participants aged 18-45 years with non-specific mid-back pain will be randomly assigned to receive either thoracic spine manipulation alone or in combination with costovertebral joint manipulation. Primary outcomes will include pain intensity measured by the Numeric Pain Rating Scale (NPRS), while secondary outcomes will involve thoracic spine range of motion measured by Bubble Inclinometer, and functional disability assessed by the Oswestry Disability Index (ODI). Statistical analysis will be performed using the statistical software IBM SPSS Statistics SPSS 25.0 for calculations. This study aims to provide evidence-based insights into the relative benefits of these manual therapy techniques, potentially informing clinical practice and enhancing treatment outcomes for patients with non-specific mid-back pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be between 18 - 45 years of age
* For this study, mid-back pain included all the following signs and symptoms:
* Sharp, shooting, or aching mid-back pain
* Mid back pain experienced during deep inspiration, sneezing, and/or coughing

Exclusion Criteria:

* Individuals who did not sign or understand the letter of informed consent
* Individuals with contraindications to manipulation in the thoracic spine (15)
* Weakened bone due to: Osteoporosis, Infection and Neoplasm

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable
Oswestry Disability Index | upto 4 weeks
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain and quality of life. Oswestry Disability Index. Purpose. used to qualify low back pain.
Bubble Inclinometer | upto 4 weeks
  A bubble inclinometer is a simple, handheld device used to measure the angle of inclination or tilt of a surface. In the context of thoracic spine assessments, it is particularly useful for quantifying the range of motion and curvature of the spine.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cibulka M, Buck J, Busta B, Neil E, Smith D, Triller R. Intra and inter observer agreement in the mobility assessment of the upper thoracic costovertebral joints. Physiother Theory Pract. 2023 Sep 2;39(9):1993-1999. doi: 10.1080/09593985.2022.2058439. Epub 2022 Mar 27. PMID 35343374
- [Background] Koivunen K, Widbom-Kolhanen S, Pernaa K, Arokoski J, Saltychev M. Reliability and validity of Oswestry Disability Index among patients undergoing lumbar spinal surgery. BMC Surg. 2024 Jan 3;24(1):13. doi: 10.1186/s12893-023-02307-w. PMID 38172794
- [Background] Kirsten Elizabeth Petrie. E. K. (2019). Costovertebral Manipulation versus Ultrasound Therapy of Rhomboid Trigger Points and a Combination Thereof in Treating Inter-scapular Pain. PQDT-Global.
- [Background] Honore M, Picchiottino M, Wedderkopp N, Leboeuf-Yde C, Gagey O. What is the effect of spinal manipulation on the pressure pain threshold in young, asymptomatic subjects? A randomized placebo-controlled trial, with a cross-over design. Chiropr Man Therap. 2020 Feb 7;28(1):6. doi: 10.1186/s12998-020-0296-1. PMID 32028982
- [Background] Masaracchio M, Kirker K, States R, Hanney WJ, Liu X, Kolber M. Thoracic spine manipulation for the management of mechanical neck pain: A systematic review and meta-analysis. PLoS One. 2019 Feb 13;14(2):e0211877. doi: 10.1371/journal.pone.0211877. eCollection 2019. PMID 30759118
- [Background] Honore M, Leboeuf-Yde C, Gagey O. The regional effect of spinal manipulation on the pressure pain threshold in asymptomatic subjects: a systematic literature review. Chiropr Man Therap. 2018 Apr 19;26:11. doi: 10.1186/s12998-018-0181-3. eCollection 2018. PMID 29713457
- [Background] Tsegay GS, Gebregergs GB, Weleslassie GG, Hailemariam TT. Effectiveness of Thoracic Spine Manipulation on the Management of Neck Pain: A Systematic Review and Meta-Analysis of Randomized Control Trials. J Pain Res. 2023 Feb 27;16:597-609. doi: 10.2147/JPR.S368910. eCollection 2023. PMID 36875686